CLINICAL TRIAL: NCT00765362
Title: Encore Mobile - Bearing Knee Study #200
Brief Title: Mobile - Bearing Knee Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Jane M. Jacob Ph.D., DJO Surgical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study 200
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Inflammatory Tissue Disorder; Osteoarthritis; Avascular Necrosis; Post-traumatic Arthritis; Secondary Arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Subjects who are candidates for a total knee replacement and meet the inclusion/exclusion criteria of the study.
  Interventions: Device: Encore Mobile-Bearing Knee

INTERVENTIONS:
Device: Encore Mobile-Bearing Knee — Used for primary total knee replacement
  Other Names: MBK

SUMMARY:
To evaluate the safety and efficacy of the Encore Mobile-Bearing Knee.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal maturity
* Less than 70 on preoperative Knee Society Score (Rating Score)
* Sufficient bone stock, as judged by radiographs, to support primary knee implant
* Patients with inflammatory tissue disorders, osteoarthritis, post-traumatic arthritis, secondary arthritis, or avascular necrosis of the femoral condyles
* Patient is not pregnant
* Primary total knee replacement
* Sufficient collateral ligaments to support device, as judged by physician during stability testing (varus/valgus and flexion/extension)
* Varus deformity <45 or valgus deformity <45 or fixed flexion deformity <90
* Patient is likely to be available for evaluation for the duration of the study
* Able and willing to sign the informed consent and follow study procedures

Exclusion Criteria:

* Skeletal immaturity
* Greater than or equal to 70 on preoperative Knee Society Score (Rating Scale)
* Previous knee surgery that has adversely affected bone stock or prior total knee replacement
* Post patellectomy
* Patient is pregnant
* Insufficient collateral ligaments, as judged by the physician
* Neurological conditions that might hinder patient's ability to follow study procedures (i.e., any that restrict physical activities such as Parkinson's Disease, Multiple Sclerosis, previous stroke which affects lower extremity).
* Varus deformity >45 or valgus deformity >45 or fixed flexion deformity >90.
* Mental conditions that may interfere with ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the patient cannot understand the informed consent process, global dementia, prior strokes that interfere the with patient's cognitive abilities, senile dementia, and Alzheimer's Disease).
* Prisoners
* Conditions that place excessive demand on the implant (i.e. Charcot's joints, muscle deficiencies, refusal to modify postoperative physical activities, skeletal immaturity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2000-01; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Carl T. Hayden VA Hospital, Phoenix, Arizona
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - S.Florida VA Found. For Research & Education, Inc., Miami, Florida
  - Great Lakes Orthopaedics, Garden City, Michigan
  - Hilton Head Island, South Carolina
  - Orthopedic Surgery Center and Sports Medicine, Edinburg, Texas
  - The Orthopedic Specialty Hospital, Murray, Utah
  - West Jordan, Utah

REFERENCES:
- See also: Sponsor company home page — http://www.djosurgical.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile Bearing Knee: Subjects who meet the inclusion/exclusion criteria and are treated and receive the Mobile Bearing Knee. The Encore Mobile Bearing Knee is intended for subjects presenting for a primary cemented knee replacement suffering from inflammatory tissue disorders, osteoarthritis, post-traumatic arthritis, secondary arthritis, or avascular necrosis of the femoral condyles. This design is indicated for subjects who have adequate, as judged by the physician, collateral ligamentous stability to support the implant.
Period: Overall Study
Arm/Group | Mobile Bearing Knee
Started | 419
Completed | 282
Not Completed | 137
Not completed — Death | 9
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 18
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 95

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Bearing Knee
Number analyzed (Participants) | 419
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 181
  >=65 years | 238
Age Continuous [Mean (Standard Deviation); unit: years] | 66.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229
  Male | 190
Region of Enrollment [Number; unit: participants]
  United States | 419

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Score Evaluation
Description: The Knee Society Score includes a knee rating and function score. This evaluation covers the knee rating score with three main parameters of pain, stability and range of motion and that flexion contracture, extension lag and misalignment should be dealt with as deductions. Thus, 100 points will be obtained by a well-aligned knee with no pain, 125 degrees of motion, and negligible anteroposterior and mediolateral instability. 50 points are allotted for pain, 25 for stability, and 25 for range of motion. Grading for KS Score: Excellent (90-100), Good (80-90), Fair (70-79) and Poor (<70).
Time Frame: 2 year
Population: Out of the 282 subjects who completed the study, only 173 were analyzed due to either the 2 year visit being completed out of window or missing data.
Measure: Mean (Standard Deviation); unit: Average Knee Rating Score
Arm/Group | Mobile Bearing Knee
Number analyzed (Participants) | 173
Average Knee Rating Score | 93.1 (9.9)

2. Primary Outcome: Knee Society Function Score
Description: The patient function score considers only walking distance and stair climbing, with deductions for walking aids. The maximum function score is obtained by a patient who can walk an unlimited distance and go up and down stairs normally. Walking ability is expressed in blocks (approximately 100 meters). Stair climbing is considered normal if the patient can ascend and descend stairs without holding a railing. A score of > or = to 60 on the function score is considered success. Minimum score = 0, maximum score = 100 with the higher the score representing a better outcome.
Time Frame: 2 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Average Knee Function Score
Arm/Group | Mobile Bearing Knee
Number analyzed (Participants) | 173
Average Knee Function Score | 89.0 (15.6)

3. Primary Outcome: Knee Society Scores Used as Success/Failure Criteria.
Description: The maximum score for each of the sections is 100 points. A score of at least 80 points on the 2-year knee assessment score was defined as a success.
Time Frame: 2 year
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants with Success
Arm/Group | Mobile Bearing Knee
Number analyzed (Participants) | 173
Percentage of Participants with Success
  Knee Society Score Success | 91
  Knee Function Score Success | 84

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of surgery through the 2 year visit.
Arm/Group | Mobile Bearing Knee
Serious Adverse Events (participants affected / at risk) | 0/419
Other Adverse Events (participants affected / at risk) | 281/419
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mobile Bearing Knee (N=419)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 12 (13)
Cancer (Immune system disorders) | 10 (10)
Degenerative Arthritis (Musculoskeletal and connective tissue disorders) | 8 (9)
Knee device clicking (Injury, poisoning and procedural complications) | 9 (9)
Edema (Blood and lymphatic system disorders) | 13 (13)
Fracture (Musculoskeletal and connective tissue disorders) | 8 (8)
Heart Complications (Cardiac disorders) | 10 (10)
Infections (Infections and infestations) | 16 (16)
Neurological disorder and numbness (Nervous system disorders) | 11 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 203 (328)
Swelling (Vascular disorders) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less